CLINICAL TRIAL: NCT00286988
Title: Topiramate for the Prophylactic Treatment of Cyclic Vomiting Syndrome in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient potential subjects
Sponsor: Monarch Medical Research (Other)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Responsible Party: Donald W Lewis, MD, Children's Specialty Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TOPMAT-EME-4001
Record Dates: First submitted 2006-02-01; First posted 2006-02-06 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2007-04

CONDITIONS: Vomiting
Keywords: Preventative; Open-Label; Safety/Efficacy
MeSH Terms: conditions — Vomiting | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
The purpose of this study is to assess the effectiveness, tolerability and safety of oral topiramate for the preventative management of Cyclic Vomiting Syndrome. It is believed that topiramate will decrease the frequency, duration and severity of attacks experienced by children and adolescents with Cyclic Vomiting Syndrome.

DETAILED DESCRIPTION:
There is very little controlled data on the preventative treatment for Cyclic Vomiting Syndrome. The existing evidence consists of small, retrospective clinical series that evaluate symptomatic responses to five medications including cyproheptadine, propranolol, amitriptyline, phenobarbital and pizotifen (n >10). These published data consist of uncontrolled or retrospective reports. In addition, varying inclusion criteria and outcomes (i.e. obtained by family recall) were used in these studies limiting the basis upon which to compare relative effectiveness.

During the prospective baseline period, the subject will maintain cyclical vomiting records in which all headache occurrences will be recorded and characterized. (Cyclical vomiting records will be maintained throughout the study). The purpose of this study is to assess the effectiveness, tolerability and safety of oral topiramate for the preventative management of Cyclic Vomiting Syndrome using a prospective design, established diagnostic criteria (ICHD 2004), and defined, objective primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Meet the2004 ICHD Criteria for Cyclical Vomiting.

  * 1 vomiting attack lasting > 24 hours duration for 3 consecutive months
* 4-12 years of age.
* If female, subjects must:

  1. be premenarchal or otherwise incapable of pregnancy, or
  2. have practiced one of the following methods of contraception for at least one month prior to study entry: hormonal contraceptives, spermicide and barrier, intrauterine device, partner sterility, or
  3. be practicing abstinence and agree to continue abstinence or to use an acceptable method of contraception (as listed above) should sexual activity commence.
* Able to take oral medication in tablet form or sprinkle form
* Subjects or their guardians must be willing and able to: a) read and comprehend written instructions, b) complete the assessment forms, c) return for regular visits, and d) adhere to medication regimens.
* Subjects (or their legally acceptable representative) must have signed an informed consent document

Exclusion Criteria

* Have taken topiramate within 14 days prior to the start of the prospective baseline period.
* Have taken certain medications for cyclical vomiting prophylaxis
* Have progressive neurological disorder or a structural disorder of the brain from birth, trauma or past infection.
* Subjects who have taken any medications for migraine prophylaxis, within 2 weeks of the start of the prospective baseline period.
* Subjects starting non-pharmacologic prophylactic approaches (e.g., acupuncture, biofeedback, chiropractic methods) within 1 month prior to Visit 1.
* Require continuing treatment with anticonvulsant therapy for a non-migraine condition.
* Significant major psychiatric disorder (e.g., major depression) or subjects receiving anti-psychotic medication.
* History of attempted suicide or suicidal tendencies.
* History of substance abuse.
* Pregnant or lactating females.
* Have clinically unstable neurological, cardiovascular, gastrointestinal, musculoskeletal, pulmonary or other disease.
* Have any disease or condition that could compromise the function of those body systems that could result in altered absorption, excess accumulation, or impaired metabolism or excretion of the test medications (e.g., abnormal renal and/or hepatic function).
* Have active liver disease.
* Have received an investigational drug or used an investigational device within 30 days of study entry.
* Employees of the investigator, study center, or sponsor (i.e., principal investigator, sub-investigator(s), study coordinators, other study staff, employees, or contractors of each), with direct involvement in the proposed study or other studies under the direction of that investigator, study center or sponsor, as well as family members of the employees or the investigator.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Reduction of cycle frequency as measured by number of days between cycles.

SECONDARY OUTCOMES:
Decreased duration of attacks (measured in hours)
Decreased intensity of attacks (0-4 point scale; none, mild, moderate, severe, excruciating)
Decreased associated symptoms (0-4 point scales; none, mild, moderate, severe, excruciating)
Nausea
Vomiting
Headache
Abdominal pain
Decreased disability
PedMidas
Missed school (days per attack)
Missed work (parent(s)) (days per attack)
Decreased use of acute therapies (e.g. anti-emetics)
Decreased emergency department visits.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Lewis, MD, Principal Investigator — Monarch Medical Research
Locations (1):
- Monarch Medical Research - Child and Adolescent Neurology, Norfolk, Virginia, United States

REFERENCES:
- [Background] CULLEN KJ, MA CDONALD WB. The periodic syndrome: its nature and prevalence. Med J Aust. 1963 Aug 3;50(2):167-73. No abstract available. PMID 14024194
- [Background] Abu-Arafeh I, Russell G. Prevalence and clinical features of abdominal migraine compared with those of migraine headache. Arch Dis Child. 1995 May;72(5):413-7. doi: 10.1136/adc.72.5.413. PMID 7618907
- See also: Click here for more information on Cyclic Vomiting Syndrome — http://www.cvsaonline.org